CLINICAL TRIAL: NCT06934824
Title: Clinical Study of Double-Endoscopic Combined With Minimally Invasive Treatment for Early Gastric Cancer at Clinical Stage T1b
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Professor, Hebei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUTURE11
Record Dates: First submitted 2025-02-09; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer Patients Undergoing Minimally Invasive Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients in group A-No lymph node metastasis, who underwent simple Double-Endoscopic Combined with local full-thickness resection.
  Interventions: Procedure: Sixty patients with early gastric cancer in stage T1bN0-1M0 were divided into Group A-N0 and Group B-N + according to the presence or absence of lymph node metastasis. When the enrolled patients und
- Group B (Experimental): Patients in group B-imaging examination showed lymph node metastasis. patients were randomly divided into Group N + a and Group N + b.
  Group N + a: Local full-thickness gastric wall and lymph nodes dissection on D1 or D1 + were performed with Double-Endoscopic Group N + b: Traditional standard surgical gastrectomy and D1 or D1 + lymph nodes dissection was performed .
  Interventions: Procedure: Sixty patients with early gastric cancer in stage T1bN0-1M0 were divided into Group A-N0 and Group B-N + according to the presence or absence of lymph node metastasis. When the enrolled patients und

INTERVENTIONS:
Procedure: Sixty patients with early gastric cancer in stage T1bN0-1M0 were divided into Group A-N0 and Group B-N + according to the presence or absence of lymph node metastasis. When the enrolled patients und — Patients in group A-No lymph node metastasis, who underwent simple Double-Endoscopic Combined with local full-thickness resection.
  Patients in group B-imaging examination showed lymph node metastasis. patients were randomly divided into Group N + a and Group N + b.
  Group N + a: Local full-thickness gastric wall and lymph nodes dissection on D1 or D1 + were performed with Double-Endoscopic Group N + b: Traditional standard surgical gastrectomy and D1 or D1 + lymph nodes dissection was performed .

SUMMARY:
For patients diagnosed with early gastric cancer involving submucosal invasion, super-ESD indications, or lymph node metastasis, a combination of preoperative endoscopic ultrasound and abdominal contrast-enhanced CT was utilized to ascertain the depth of tumor invasion and to identify any suspicious metastatic lymph nodes in the vicinity of the stomach. Subsequently, a local full-thickness resection, coupled with or followed by individualized precise lymph node dissection, was conducted to fulfill the following objectives: ① To investigate the safety, feasibility, and efficacy of local resection for patients meeting super-ESD criteria; ② To offer a clinical foundation for the individualized and precise lymph node dissection treatment of early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old;
2. Endoscopic pathological diagnosis: adenocarcinoma;
3. Enhanced abdominal CT combined with endoscopic ultrasound clinical staging: T1bN0-1M0.
4. Has not received other treatment;
5. No other serious comorbidities;
6. Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. History of previous abdominal surgery
3. History of other previous malignancies
4. Can patients with severe heart, lung, brain diseases tolerate surgical treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence | Within 2 years

SECONDARY OUTCOMES:
The operation time, complications and hospital stay were recorded | 30 days

IPD SHARING:
Plan to Share IPD: Undecided